CLINICAL TRIAL: NCT04986241
Title: Retrospective Study of the Association of Statins on Cardiorespiratory Fitness and Exercise Adaptation: Database of the Cardiovascular Rehabilitation and Exercise Physiology Department of Heart Institute (InCor)
Brief Title: The Association of Statins on Cardiorespiratory Fitness and Exercise Adaptation
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CardioRehab Bank Study
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2022-10

CONDITIONS: Statin Adverse Reaction
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Sedentary Heart Failure with Reduced Ejection Fraction Without Statin: Sedentary Heart Failure with Reduced Ejection Fraction determined by echocardiogram; Without statin in the last 6 months.
  Interventions: Other: Sedentary
- Sedentary Heart Failure with Reduced Ejection Fraction With Statin: Sedentary Heart Failure with Reduced Ejection Fraction determined by echocardiogram; With current use of statin.
  Interventions: Drug: Statin; Other: Sedentary
- Physically active Heart Failure with Reduced Ejection Fraction Without Statin: Physically active Heart Failure with Reduced Ejection Fraction determined by echocardiogram; Without statin in the last 6 months.
  Interventions: Other: Physical activity
- Physically active Heart Failure with Reduced Ejection Fraction With Statin: Physically active Heart Failure with Reduced Ejection Fraction determined by echocardiogram; With current use of statin.
  Interventions: Drug: Statin; Other: Physical activity
- Healthy sedentary Without Statin: Sedentary and healthy participant without use of statin; Without statin in the last 6 months.
  Interventions: Other: Sedentary
- Healthy sedentary With Statin: Participant with dyslipidemia and sedentary with current use of statin.
  Interventions: Drug: Statin; Other: Sedentary
- Healthy physically active Without Statin: Healthy, physically active participant without use of statin; Without statin in the last 6 months.
  Interventions: Other: Physical activity
- Healthy physically active With Statin: Participant with dyslipidemia and physically active with current use of statin.
  Interventions: Drug: Statin; Other: Physical activity

INTERVENTIONS:
Drug: Statin — Chronic use of statin prescribed previously by the assistant physician.
  Other Names: 3-hydroxy-3-methyl-glutaryl-coenzyme A reductase inhibitor
  Groups: Healthy physically active With Statin; Healthy sedentary With Statin; Physically active Heart Failure with Reduced Ejection Fraction With Statin; Sedentary Heart Failure with Reduced Ejection Fraction With Statin
Other: Physical activity — Physically active participants
  Other Names: Physical exercise
  Groups: Healthy physically active With Statin; Healthy physically active Without Statin; Physically active Heart Failure with Reduced Ejection Fraction With Statin; Physically active Heart Failure with Reduced Ejection Fraction Without Statin
Other: Sedentary — Physically inactive or sedentary participants.
  Other Names: Physical inactivity
  Groups: Healthy sedentary With Statin; Healthy sedentary Without Statin; Sedentary Heart Failure with Reduced Ejection Fraction With Statin; Sedentary Heart Failure with Reduced Ejection Fraction Without Statin

SUMMARY:
Statins are part of one of the largest groups of drugs prescribed worldwide used in the treatment of dyslipidemia. Despite the good therapeutic results of statins and their good tolerance on the part of patients, some adverse effects may occur during treatment. In skeletal muscle, statins can lead to mitochondrial dysfunction characterized by decreased adenosine triphosphate production, decreased oxidative phosphorylation capacity, increased concentration of reactive oxygen species, and decreased mitochondrial biogenesis.

Cardiorespiratory fitness is a physiological indicator that corresponds to the integration of the cardiovascular, pulmonary, muscular, and cellular (mitochondria) systems in capturing, transporting and using oxygen, commonly expressed as the maximum oxygen consumption. Several studies show a strong association of lower cardiorespiratory capacity with an increased risk of mortality from cardiovascular disease and mortality from all causes.

Combining the use of statins with lifestyle changes has been suggested in many medical guidelines. Physical exercise plays a fundamental role in improving cardiorespiratory fitness and controlling dyslipidemia. However, some studies suggest that the association of statin with physical training can negatively influence the adaptation and improvement of cardiorespiratory capacity. On the other hand, some studies show that the combination of statin and physical exercise does not negatively interfere with the maximum oxygen consumption.

To determine the impact of statins on cardiorespiratory fitness and adaptation to physical exercise, the investigators will use the database of the Cardiovascular Rehabilitation and Exercise Physiology Department at Heart Institute (Sao Paulo, Brazil), which currently has 33,804 maximal cardiopulmonary exercise tests. This large database, which is the gold standard of cardiorespiratory capacity (maximum oxygen consumption), will be used retrospectively with relevant information and a huge number of participants.

Therefore, the aim of this study will be to explore a large database to assess the effect of the use of statins and their relationship with cardiorespiratory capacity in physically active and sedentary individuals (with and without heart failure).

DETAILED DESCRIPTION:
The investigators will use the database of the Cardiovascular Rehabilitation and Exercise Physiology Department at Heart Institute (Sao Paulo, Brazil) in an exploratory manner. The investigators will use filters to perform different analyzes and sub-analyses with different groups of patients. The investigators aimed to compare patients using statins and healthy controls (not using medications). The analysis strategy will be as following: 1) physically active and sedentary patients with normal cardiac function using statins and peak oxygen consumption (peak VO2); 2) physically active and sedentary patients with cardiac dysfunction (heart failure) using statins and peak VO2; 3) comparison between the hydrophilic and lipophilic classes of statins; 4) comparison between men and women; 5) retrospective information on clinical and laboratory variables and 6) test information on cardiorespiratory capacity and several variables associated with the mortality outcome.

The participants underwent cardiopulmonary exercise testing on a treadmill or bike (SensorMedics - Vmax Analyzer Assembly, Encore 29S) following a ramp protocol with constant load increase until exhaustion. Cardiorespiratory capacity will be determined by peak VO2, assessed at maximum exercise intensity, with a respiratory exchange ratio >1.10.

ELIGIBILITY:
Inclusion Criteria:

* Maximal Cardiopulmonary Test on treadmill or bike.
* Test considered maximum from the metabolic point of view (Respiratory Quotient >1.10).

Exclusion Criteria:

* Incomplete patient data.
* Incomplete exam data.
* Chronic obstructive pulmonary disease
* Diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study are patients admitted in the Cardiovascular Rehabilitation and Exercise Physiology Department at Heart Institute Hospital (Sao Paulo, Brazil) for a cardiopulmonary exercise test.
Sampling Method: Probability Sample
Enrollment: 18557 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | From 1998 to 2017
  To determine whether the use of statins impairs the adaptation of the cardiorespiratory fitness in physically active individuals, with and without left ventricular dysfunction (heart failure), when compared with a matched sedentary control group.

SECONDARY OUTCOMES:
Types of statins in Cardiorespiratory Fitness | From 1998 to 2017
  To determine whether the type of statins (lipophilic or hydrophilic) has any adverse effect on the cardiorespiratory fitness in physically active individuals, with and without left ventricular dysfunction (heart failure), when compared with a matched sedentary control group.
Sex differences | From 1998 to 2017
  To determine whether sex (men and women) is associated with statins and cardiorespiratory fitness impairment.
Cardiovascular mortality | From 1998 to 2017
  To determine the association of functional capacity and cardiorespiratory fitness with cardiovascular mortality.
All-cause mortality | From 1998 to 2017
  To determine the association of functional capacity and cardiorespiratory fitness with all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo R dos Santo, PhD, Principal Investigator — Instituto do Coracao (InCor)
Locations (1):
- Marcelo Rodrigues dos Santos, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No